CLINICAL TRIAL: NCT00202514
Title: Placebo Controlled Trial of Depakote ER in Alcohol Dependent Patients With Mood and/or Anxiety Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Abbott (Industry)
Responsible Party: Joseph P. Reoux, MD, Seattle Institute for Biomedical and Clinical Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R&D protocol #: RDIS 0009
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Alcoholism; Alcohol Related Disorders; Mood Disorders
Keywords: alcoholism; alcohol related disorders; mood disorders; anticonvulsants; divalproex sodium
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: divalproex sodium extended release

SUMMARY:
The purpose of this study is to test the safety and effectiveness of an extended release form of a medication called divalproex sodium (Depakote ER) for the treatment of people with alcohol dependence who have mood and/or anxiety symptoms. This medication has helped reduce symptoms of acute alcohol withdrawal as well as stabilize mood symptoms in bipolar disorder and other mental health disorders. This study will test the hypothesis that divalproex sodium will help reduce mood and anxiety symptoms during early abstinence from alcohol and in turn reduce relapse and craving for alcohol.

DETAILED DESCRIPTION:
Alcohol dependence afflicts 14 million individuals in the U.S. The alcohol related costs to society are enormous and alcohol dependence is a significant public health problem. Although pharmacotherapy for the treatment of alcohol dependence and relapse prevention has expanded, the identification of evidence based treatment strategies is of critical importance. Anticonvulsants, including the divalproex sodium (DVP) formulation of valproate, have established effectiveness for mood disorders, and therapeutic response of mood and anxiety symptoms to DVP has been demonstrated in a number of psychiatric conditions. While DVP has been demonstrated as a treatment option for the acute alcohol withdrawal syndrome, a clear treatment effect has not been found in studies examining DVP for ongoing relapse prevention in alcohol dependence. These latter studies had limited power and excluded subjects with co-morbid mood and anxiety disorders, individuals who may, by extension of the former studies, show the greatest response to treatment with DVP. Despite the exclusion of subjects with mood and anxiety disorders, alcohol dependent individuals treated with DVP compared to placebo showed greater improvement in irritability and a trend toward greater decreases on measures of impulsivity and aggression. A strategy integrating the above findings would target treatment with DVP more specifically to alcohol dependent individuals with mood and anxiety disturbances.

This randomized, double-blind clinical trial will examine the effectiveness of extended release DVP (Depakote-ER) in the treatment of co-morbid mood and anxiety disturbance in alcohol dependent subjects. The primary hypothesis is that subjects treated with Depakote-ER will have significantly lower scores on the Symptom Checklist (SCL-90-R) than will placebo treated subjects over the course of the study. Secondary hypotheses include: 1) Compared to placebo treated subjects, subjects treated with Depakote-ER will demonstrate significantly lower scores on additional measures of depression, anxiety, and irritability, 2) will have fewer alcohol use days and fewer drinks per drinking day, and 3) will evidence better retention in alcohol dependence treatment.

Eligible subjects will complete baseline assessments and a 7-day run on Depakote-ER prior to randomization. After the 7-day baseline period and run in with Depakote-ER, subjects will be randomized and then transition to either 12 weeks of Depakote-ER or placebo, to begin upon completion of the 7-day run-in baseline period. Valproic acid level obtained at the end of the baseline period will be used to adjust the dose of Depakote-ER (or matched placebo) as needed to target a valproic level of 70-120 ug/ml. Dose increase, if needed, will occur with the study medication dispensed at the next follow up visit (scheduled for the end of the 1st week of active study medication or placebo). Subjects with valproic acid levels > 120 ug/ml at the end of the baseline period will be contacted as soon as possible and instructed to decrease their dose of Depakote-ER (or matched placebo) accordingly. Subjects randomized to the placebo condition will receive a placebo matched in number and appearance to the dosage of Depakote-ER prescribed during the 7-day baseline period. If needed, the number of placebo pills will be adjusted to match the change in the Depakote-ER dosage determined necessary based on the valproic acid level obtained at the end of the 7-day baseline period.

Duration of Subject Participation: Subjects will receive either divalproex sodium extended release (Depakote-ER) or matched placebo for 12 weeks. Subjects will continue to receive other "treatment as usual" within the Addiction Treatment Center in accordance with their ongoing clinical program treatment plan. The standard expectation within the context of treatment as usual is for at least 6 months of treatment involvement. A limited number of psychotropic medications will be allowed during the study. A benzodiazepine (usually chlordiazepoxide or lorazepam, in accordance with standard practice and generally given in an as needed symptom triggered manner) can be prescribed during the acute detoxification period (first 7 days). Hydroxyzine can be prescribed PRN for anxiety, and zolpidem PRN (not to exceed 5 nights per week) for insomnia, throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant or nursing female age 18 to 65 years old.
2. Females of childbearing potential must agree to practice an acceptable form of birth control during the time enrolled in the study.
3. Diagnosis of DSM-IV alcohol dependence (DSM-IV checklist).
4. Sub-syndromal mood and/or anxiety symptoms (threshold score of 1 standard deviation above the mean for non-psychiatric population on the anxiety, depression, hostility, or global severity subscales of the SCL-90).
5. Subjects must be able to understand and sign an informed consent approved by the center's Institutional Review Board.

Exclusion Criteria:

1. Opioid dependence as the primary substance diagnosis.
2. Clearly established non-substance related psychiatric disorder determined by administration of the Structured Clinical Interview for DSM-IV (SCID-IV) requiring immediate medication treatment.
3. Concurrent need for ongoing treatment with a benzodiazepine, anticonvulsants, or medications with significant drug-drug interaction with DVP.
4. Severe liver disease (ascites, jaundice, encephalopathy) suggested by physical exam.
5. AST or ALT > 200 U/L; total bilirubin > 2.5 mg/dl.
6. PT > 1.5X normal.
7. Platelet count < 100,000/cubic mm, or WBC < 3,000/cubic mm.
8. Pancreatitis (clinical signs and symptoms, not solely based on blood tests).
9. Known allergy to DVP or valproic acid.
10. Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
mood and anxiety symptoms over time [SCL-90-R (Symptom Check List)].

SECONDARY OUTCOMES:
scores on additional measures of depression (Ham-D),
scores on additional measures of anxiety (Ham-A),
scores on additional measures of irritability (AIAQ),
Alcohol and other drug consumption (timeline followback),
urine toxicology,
Alcohol craving (Obsessive-Compulsive Drinking Scale),
medication side effects,
sleep diary,
concomitant medication use,

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Reoux, MD, Principal Investigator — Veterans Affairs and University of Washington
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Background] Brady KT, Myrick H, Henderson S, Coffey SF. The use of divalproex in alcohol relapse prevention: a pilot study. Drug Alcohol Depend. 2002 Aug 1;67(3):323-30. doi: 10.1016/s0376-8716(02)00105-9. PMID 12127203
- [Background] Hertzman M. Divalproex sodium to treat concomitant substance abuse and mood disorders. J Subst Abuse Treat. 2000 Jun;18(4):371-2. doi: 10.1016/s0740-5472(99)00080-x. PMID 10812311
- [Background] Reoux JP, Saxon AJ, Malte CA, Baer JS, Sloan KL. Divalproex sodium in alcohol withdrawal: a randomized double-blind placebo-controlled clinical trial. Alcohol Clin Exp Res. 2001 Sep;25(9):1324-9. PMID 11584152